CLINICAL TRIAL: NCT00827229
Title: Evaluation of Laborpro - a New Device for the Assessment of Progress of Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trig Medical Inc (Industry)
Responsible Party: Yoav paltieli CEO, Trigmedical
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CLP 019/2008CTIL
Record Dates: First submitted 2009-01-21; First posted 2009-01-22 (Estimated); Last update posted 2009-01-22 (Estimated); Status verified 2009-01

CONDITIONS: Labor
Keywords: Active labor; Term pregnancy; Vertex presentation; Single fetus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LaborPro, active Labor, Vaginal Examination (Other)
  Interventions: Device: Labor Monitor

INTERVENTIONS:
Device: Labor Monitor

SUMMARY:
A clinical study was conducted to demonstrate the accuracy of the LaborPro System in measuring fetal head station (from the pelvic inlet), cervical dilatation, and fetal head position against manual/digital examination. The LaborPro obtained device values was compared to measurements gathered within 15 minutes by manual/digital examination performed by two independent physicians. The study was a non significant risk (NSR) device study.

DETAILED DESCRIPTION:
Objective The purpose of the study was to evaluate the accuracy of LaborPro fetal head station, fetal head position, and cervical dilatation measurements as compared to manual/digital examinations and to demonstrate that the LaborPro System is safe.

Methods and Procedures The study population included of women admitted to either Maimonides Medical Center (NY, USA) or Bnai Zion Medical Center (Haifa, Israel) in the active phase of labor, with singleton pregnancy and vertex presentation. One hundred and ten (110) subjects were enrolled in the study. Two subjects were excluded from the study as one from Bnai Zion Medical Center had a system malfunction (PC failure) and one subject from Maimonides Medical Center changed her mind and refused to participate in the study. Sixty Seven (67) subjects (62%) were enrolled at Maimonides Medical Center and forty one (41) subjects (38%) were enrolled at Bnai Zion Medical Center. Subject's mean age was 28.2 years (ranging from 15.8 years to 39.5).

Each subject was examined and in cases in which the first exam (according to blinded physician assessment) was at an early labor stage (cervical dilatation < 3 cm), a second examination interval of at least 2 hours after the first one was recorded. In cases where the first examination was performed at a more advanced labor stages (cervical dilatation > 3 cm), a second examination interval was recorded at least 1 hour after the first one. Each set of examinations (LaborPro and two independent practitioners) of station, position and cervical dilatation was completed within 15 minutes. The two independent physicians were blinded to each other's results and to the LaborPro results. If labor duration enabled further examination, two to three sets of tests were performed for each subject. During labor, the attending physician, a midwife or nurse conducted manual trans-vaginal digital evaluations (TVDEs) according to standard practice with respect to frequency and method.

During the manual TVDE, the clinician used the LaborPro finger sensor so that simultaneous LaborPro measurements of fetal head station finger tip (HSFT) and cervical dilatation (CDFT) were recorded. A trained ultrasonographer (physician, midwife or technician) also performed an ultrasound examination to yield the LaborPro data for measurements of head position (HP) and the head station (HSUS) with respect to BPD vs. Pelvic Inlet or with respect to fetal scalp tip vs. Pelvic Inlet.

Study Endpoints Primary Endpoint The primary efficacy endpoints of the study are average differences between measurements of Head Station (HS) and Cervical Dilatation (CD) made by the device (LaborPro) and by TVDEs.

Secondary Endpoint The secondary efficacy endpoint is the degree of agreement between the Fetal Head Position (HP) measured by LaborPro versus the one measured by TVDE.

In summary, the labor parameters as measured by LaborPro compared to the gold-standard physicians' assessment result in an accurate representation of fetal head station (calculated from the pelvic inlet), cervical dilatation, and fetal head position. It therefore can be concluded that the LaborPro provides a clinically and statistically adequate estimate of the fetal head station (calculated from the pelvic inlet), fetal head position, and cervical dilatation. The safety profile of the LaborPro non invasive system is also demonstrated by the non occurrence of any device related adverse event.

ELIGIBILITY:
Inclusion Criteria:

* Active phase of labor
* Singleton pregnancy (as diagnosed by ultrasound)
* Cephalic presentation

Exclusion Criteria:

* Known or suspected disease of mother or fetus from among the following:
* Positive HIV testing
* Positive Hepatitis B Surface Antigen testing
* Active Genital Herpes Simplex
* Coagulation disorders
* Fetal distress
* Inability to provide informed consent or comply with study protocol
* Abnormal placentation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2007-01; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)